CLINICAL TRIAL: NCT01499485
Title: Effects of Acetazolamide on the Duration of Mechanical Ventilation in Patients With Metabolic Alkalosis. Phase III Multicenter Double-blinded Clinical Trial.
Brief Title: Treatment of Metabolic Alkalosis With Acetazolamide. Effect on the Length of Mechanical Ventilation.
Acronym: TRAMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Gemma Rialp, MD; PhD, Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRAMA study
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome; Metabolic Alkalosis
Keywords: Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome; Alkalosis; Respiration, Artificial; Acetazolamide; Intensive care; Adult
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome; Alkalosis; Respiratory Aspiration | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Experimental)
  Interventions: Drug: Acetazolamide
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Daily morning ABGA:
  * If actual bicarbonate > 26 mmol/L and pH > 7.35: administration of enteral capsule of acetazolamide 500 mg .
  * If actual bicarbonate > 26 mmol/L and pH <= 7.35, increase minute ventilation to reach pH > 7.35 and then administer enteral capsule of acetazolamide 500 mg.
  * If actual bicarbonate <= 26 mmol/L: omit treatment that day.
  Other Names: Edemox
  Arms: Acetazolamide
Drug: Placebo — Daily morning ABGA:
  * If actual bicarbonate > 26 mmol/L and pH > 7.35: administration of enteral capsule of placebo.
  * If actual bicarbonate > 26 mmol/L and pH <= 7.35, increase minute ventilation to reach pH > 7.35 and then administer enteral capsule of placebo.
  * If actual bicarbonate <= 26 mmol/L: omit treatment that day.
  Arms: placebo

SUMMARY:
The purpose of this study is to analyze whether the treatment of metabolic alkalosis with acetazolamide in intubated patients with chronic obstructive pulmonary disease (COPD) or with obesity hypoventilation syndrome (OHS) reduces the length of mechanical ventilation (MV).

DETAILED DESCRIPTION:
Metabolic alkalosis (MA) may reduce central respiratory drive, cardiac output and worsen oxygenation, leading to a delay in weaning from MV. Acetazolamide is a carbonic anhydrase inhibitor that is able to correct MA and to stimulate respiratory drive. There is a paucity of studies on the outcome of patients with MA under MV treated with acetazolamide.

The primary objective of our study is to analyze whether the treatment of MA with acetazolamide in intubated patients with COPD or with OHS reduces the length of MV, reduces the length of ICU stay or ICU mortality. Complications associated with acetazolamide treatment will be also analyzed.

Phase III double-blinded trial, with COPD or OHS patients under MV who have pH > 7,35 and bicarbonate > 28 mEq/L. Patients will be randomized to receive 500 mg of acetazolamide or placebo. According to arterial blood gas analysis (ABGA) values treatment administration will be evaluated daily until extubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD or obesity hypoventilation syndrome on invasive mechanical ventilation during less than 72 h with metabolic alkalosis, defined as a pH > 7.35 and actual bicarbonate > 28 mmol/L, and with potassium plasmatic levels >= 4 mEq/L.

Exclusion Criteria:

* Postoperative patients.
* Previous psychiatric disease.
* Epilepsy.
* Pregnancy.
* Hepatic cirrhosis.
* Sulfonamide or acetazolamide allergy.
* Plasmatic creatinine > 2.5 mg/dL or creatinine clearance < 20 mL/min or continuous renal replacement techniques.
* Intolerance to enteral feeding.
* Administration in the previous 72 h of bicarbonate or acetazolamide.
* Terminal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Length of mechanical ventilation | From intubation date to extubation date, an expected average of 1 week

SECONDARY OUTCOMES:
Length of intensive care unit stay | The duration of ICU stay, an expected average less than 2 weeks
All cause hospital mortality | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Alive or dead status will be recorded at the end of hospital stay
Complications associated to the treatment | During the mechanical ventilation period, an expected average of 1 week
  Plasma and urine analysis will be performed to detect alteration in electrolites or renal function.

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital de Manacor, Manacor, Balearic Islands
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Fundació Hospital Asil de Granollers, Granollers, Barcelona
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid

REFERENCES:
- [Background] Faisy C, Mokline A, Sanchez O, Tadie JM, Fagon JY. Effectiveness of acetazolamide for reversal of metabolic alkalosis in weaning COPD patients from mechanical ventilation. Intensive Care Med. 2010 May;36(5):859-63. doi: 10.1007/s00134-010-1795-7. Epub 2010 Mar 9. PMID 20217045
- [Background] Raurich JM, Rialp G, Ibanez J, Llompart-Pou JA, Ayestaran I. Hypercapnic respiratory failure in obesity-hypoventilation syndrome: CO(2) response and acetazolamide treatment effects. Respir Care. 2010 Nov;55(11):1442-8. PMID 20979670
- [Background] Mazur JE, Devlin JW, Peters MJ, Jankowski MA, Iannuzzi MC, Zarowitz BJ. Single versus multiple doses of acetazolamide for metabolic alkalosis in critically ill medical patients: a randomized, double-blind trial. Crit Care Med. 1999 Jul;27(7):1257-61. doi: 10.1097/00003246-199907000-00004. PMID 10446816
- [Background] Banga A, Khilnani GC. Post-hypercapnic alkalosis is associated with ventilator dependence and increased ICU stay. COPD. 2009 Dec;6(6):437-40. doi: 10.3109/15412550903341448. PMID 19938966
- [Background] Moviat M, Pickkers P, van der Voort PH, van der Hoeven JG. Acetazolamide-mediated decrease in strong ion difference accounts for the correction of metabolic alkalosis in critically ill patients. Crit Care. 2006 Feb;10(1):R14. doi: 10.1186/cc3970. PMID 16420662
- [Derived] Rialp Cervera G, Raurich Puigdevall JM, Moran Chorro I, Martin Delgado MC, Heras la Calle G, Mas Serra A, Vallverdu Perapoch I. Effects of early administration of acetazolamide on the duration of mechanical ventilation in patients with chronic obstructive pulmonary disease or obesity-hypoventilation syndrome with metabolic alkalosis. A randomized trial. Pulm Pharmacol Ther. 2017 Jun;44:30-37. doi: 10.1016/j.pupt.2017.03.002. Epub 2017 Mar 7. PMID 28286047